CLINICAL TRIAL: NCT01962233
Title: Safety and Efficacy Investigation of Patients With Hypoxic Ischemic Encephalopathy by Transplantation of Umbilical Cord Derived Mesenchymal Stem Cells
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells Therapy in Hypoxic Ischemic Encephalopathy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of Cell Thearpy Center, the First Hospital of HeibeiMU, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12276102D-Neurologic Disorder
Record Dates: First submitted 2013-09-11; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-09

CONDITIONS: Hypoxic Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cells (Experimental): Umbilical Cord Derived Mesenchymal Stem Cells at a dose of 100-800 million by intravenous infusion
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — Procedure: On the basis of conventional therapy, at the same time, selected patients were given by intravenous infusion of umbilical cord blood stem cells 100-800 million. All patients before treatment, after treatment for 15days, 90days and 180 days were evaluated respectively the curative effect.
  Intravenous infusion of umbilical cord derived mesenchymal stem cells

SUMMARY:
This study is to evaluate the safety and efficacy of Umbilical Cord Derived Mesenchymal Stem Cells transplantation in hypoxic ischemic encephalopathy.

DETAILED DESCRIPTION:
To date,hypoxic ischemic encephalopathy is refractory, including after carbon monoxide poisoning, cardiopulmonary resuscitation,hemorrhagic shock and cerebral infarction etc. We used Mesenchymal Stem Cells via portal vein infusion method to treat hypoxic ischemic encephalopathy. With different durations of follow-up, we cleared therapeutic effect, the quality of life and prognostic implications of the cord blood stem cell infusion on hypoxic ischemic encephalopathy, and evaluated the adverse reactions, through the neurological function score (NIHSS，Barthel Index), cognitive score (MoCA, MMSE),and the international uniform Parkinson Rating Scale score (UPDRS). Here, we seek new means for the treatment of hypoxic ischemic encephalopathy, and provide the basis for clinical for further application of umbilical cord blood derived Mesenchymal stem cells.

On the basis of conventional therapy, at the same time, selected patients were given by intravenous infusion of umbilical cord blood stem cells 100-800 million. All patients before treatment, after treatment for 15days, 90days and 180 days were evaluated respectively the curative effect. The neurological function score (NIHSS score, Barthel Index) was observed in patients with the ability to live independently and prognosis; MoCA, MMSE were used in the evaluation of cognitive function ；UPDRS was used in the evaluation of extrapyramidal tract function.

ELIGIBILITY:
Inclusion Criteria:

Patients are screened foe enrollment in the study if both clinal signs and laboratory tests meet the diagnosis standards recommended by International Classification of Diseases-10 about hypoxic ischemic encephalopathy.

Exclusion Criteria:

Exclusion Criteria are any clinically significant diseases in liver,kidney,and heart. additional exclusion criteria are no pregnancy,no immunosuppressive medication, no tumor, no viral diseases or diseases associated with immunodeficiency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) scores. | 180 days
  The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42 (dead).

SECONDARY OUTCOMES:
The Barthel Index | before treatment and post cell transplantation:15,90,180 days
  The Barthel Index measures 10 activities of daily living and mobility. A score of 100 is best (able to live at home with a degree of independence), 0 is worst.
The Mini-Mental State Examination (MMSE) | before treatment and post cell transplantation:15,90,180 days
  The Mini-Mental State Examination (MMSE) is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function.
The Montreal Cognitive Assessment(MoCA) | before treatment and post cell transplantation:15,90,180 days
  The Montreal Cognitive Assessment(MoCA) is a brief 30-point screening instrument that was developed and validated to identify subjects with mild cognitive impairment. 30 is the maximum score, with a score of 26 or higher considered normal and below 26 indicative of Mild Cognitive Impairment.
Unified Parkinson's Disease Rating Scale (UPDRS) | before treatment and post cell transplantation:15,90,180 days.
  The UPDRS score has 4 components. Part I assesses mentation; Part II assesses activities of daily living; Part III assesses motor abilities; Part IV assesses complications of therapy. A total of 44 items are included in Parts I-III. Each item will receive a score ranging from 0 to 4 where 0 represents the absence of impairment and 4 represents the highest degree of impairment. Part IV contains 11 items, 4 of these items are scored 0-4 in the same manner, and 7 are scored 0-1, with 0 indicating the absence of impairment and 1 indicating the presence of impairment. Total UPDRS score represents the sum of these items in Parts I-IV. A total of 199 points are possible. 199 represents the worst (total) disability), 0--no disability.
adverse reaction | post cell transplantation:15,90,180 days
  adverse reaction include temperature changes,the change of blood pressure,anaphylaxis,seizure,renal dysfunction,or hepatic injury by monitoring blood routine, urinalysis, ALT,AST,Urea,Crea and electrocardiogram etc.

CONTACTS AND LOCATIONS:
Overall Officials: Baoyong Yan, Doctor, Study Chair — The First Hospital of Hebei Medical University; Ping Gu, Doctor, Study Director — The First Hospital of Hebei Medical University; Yanyong Wang, Doctor, Principal Investigator — The First Hospital of Hebei Medical University; Lina Zhang, Master, Principal Investigator — The First Hospital of Hebei Medical University; Jun Zhang, Master, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China